CLINICAL TRIAL: NCT01067391
Title: A Randomized, Double-blind, Placebo-controlled Cross-over Trial Assessing the Effect of Tadalafil (Cialis) on the Cardiovascular System in Men With Complete Spinal Cord Injury (SCI) at or Above the Sixth Thoracic Level
Brief Title: Effect of Tadalafil (Cialis) on the Cardiovascular System of Spinal Cord Injury (SCI) Males
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other); Rick Hansen Foundation (Other)
Responsible Party: Principal Investigator, Dr. Karen Ethans, Director, Spinal Cord Injury Rehabilitation Program, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cialis 2009
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Hypotension; Spinal Cord Injury
Keywords: Hypotension in SCI males; Erectile Dysfunction
MeSH Terms: conditions — Hypotension; Spinal Cord Injuries; Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tadalafil 20 mg (Active Comparator): Oral study medication to be administered once to each participant
  Interventions: Drug: tadalafil
- placebo (Placebo Comparator): oral study medication to be administered once to each study participant
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tadalafil — 20 mg tablet, administered once per study protocol
  Other Names: Cialis
  Arms: tadalafil 20 mg
Drug: placebo — placebo tablet administered once per study protocol
  Arms: placebo

SUMMARY:
To address the effect of tadalafil (Cialis) on the cardiovascular system of men with complete spinal cord injury at T-6 and above. The hypothesis is that tadalafil will cause significant hypotension in people with tetraplegia.

DETAILED DESCRIPTION:
Tadalafil is a long-acting PDE-5 inhibitor, used to treat erectile dysfunction (ED). ED is a common issue for males with spinal cord injury (SCI).Patients with SCI are at risk of developing orthostatic hypotension, especially those with an injury at or above the T-6 level.An earlier study of the shorter-acting PDE-5 inhibitor sildenafil (Viagra) revealed that it can cause orthostatic hypotension, tachycardia and dizziness after administration in the SCI population, and suggested that caution should be used in prescribing sildenafil in this population, as blood pressure can drop significantly. There is potential for the significant hypotension seen with the short-acting medications to be much more problematic with the longer-acting tadalafil.

The study will be a prospective, randomized, double-blind, placebo-controlled cross-over design. This will be done by comparing the effects of administering tadalafil 20 mg and placebo on blood pressure (lying and sitting), and heart rate (lying and sitting). These measurements will be taken in the clinic setting prior to dosing, then repeated hourly for the first two hours post-dose, and again at four hours post-dose. The patient will repeat the measurements at home using an automated blood pressure apparatus at 12, 22,29 and 36 hours post-dose.In addition, the patient will record perceived dizziness on a visual analog scale ecah time the BP and HR are recorded.

ELIGIBILITY:
Inclusion Criteria:

* males 18 to 70 years old, with complete spinal cord injury (ASIA-A) between C-4 and T-6
* minimum 6 months post-injury

Exclusion Criteria:

* diabetic
* taking nitroglycerin
* ischemic heart disease or significantly abnormal EKG
* lower motor neuron dysfunction
* heroin or cocaine use
* history of adverse reaction to tadalafil or any other PDE-5 inhibitor
* any condition that may put the subject at risk, confound the study results, or interfere significantly with subject's ability to participate in the study
* have used any other (PDE-5) medications within 1 week of study medication administration

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Supine and sitting blood pressure and heart rate (HR), as well as perceived dizziness upon sitting up. | Pre-dose, 1 hour, 2, 4, 12, 22, 29 and 36 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Karen D. Ethans, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre Rehabilitation Hospital, Winnipeg, Manitoba, Canada